CLINICAL TRIAL: NCT03357952
Title: A Randomized, Open-label, Multicenter, Multiphase Study of JNJ-63723283, an Anti-PD-1 Monoclonal Antibody, Administered in Combination With Daratumumab, Compared With Daratumumab Alone in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of JNJ-63723283, an Anti-programmed Death-1 Monoclonal Antibody, Administered in Combination With Daratumumab, Compared With Daratumumab Alone in Participants With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108381; 2017-002611-34 (EudraCT Number); 54767414MMY2036 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-11-13; First posted 2017-11-30 (Actual); Results first posted 2019-11-12 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part 1: JNJ-63723283 + Daratumumab (Experimental): Participants in Safety Run-in cohort will receive daratumumab IV and JNJ-63723283 IV for 1 cycle (28 days). Participants will continue to receive study treatment until confirmed disease progression, unacceptable toxicity, or any other treatment discontinuation criteria are met. Participants who were previously receiving JNJ-283 plus daratumumab have the opportunity to continue daratumumab therapy alone.
  Interventions: Drug: Daratumumab; Drug: JNJ-63723283
- Part 2 and Part 3: Daratumumab/ JNJ-63723283 + Daratumumab (Experimental): Participants in Treatment Arm A will receive daratumumab IV and in Treatment Arm B will receive daratumumab IV and JNJ-63723283 IV for cycles of 28 days each. All participants will continue to receive study treatment until confirmed disease progression, unacceptable toxicity, or any other treatment discontinuation criteria are met. Participants who were previously receiving JNJ-283 plus daratumumab have the opportunity to continue daratumumab therapy alone.
  Interventions: Drug: Daratumumab; Drug: JNJ-63723283

INTERVENTIONS:
Drug: Daratumumab — Participants will receive daratumumab 16 milligram per kilogram (mg/kg) intravenously (IV) once every week for 8 weeks (Weeks 1 to 8); then once every other week for 16 weeks (Weeks 9 to 24); then once every 4 weeks (Week 25 onwards).
  Other Names: JNJ-54767414
Drug: JNJ-63723283 — Participants will receive JNJ-63723283 240 mg IV during Week 1 on Cycle 1 Day 2, Cycle 1 Day 15, then every 2 weeks thereafter.

SUMMARY:
The main purpose of this study is to assess the safety of the combination of JNJ-63723283 and daratumumab (Part 1); to compare the overall response rate (ORR) in participants treated with JNJ-63723283 in combination with daratumumab versus daratumumab alone (Part 2); and to compare progression-free survival (PFS) in participants treated with JNJ-63723283 in combination with daratumumab versus daratumumab alone (Part 3).

DETAILED DESCRIPTION:
This is a multi-phase study of JNJ-63723283 in combination with daratumumab compared with daratumumab alone in participants with multiple myeloma who have received at least 3 prior lines of therapy including a proteasome inhibitor (PI) and an immunomodulatory agent (IMiD) or whose disease is double refractory to both a PI and an IMiD. The study consists of Screening Phase (procedures performed within 28 days before enrollment), Open-Label Treatment Phase (with End-of-Treatment Visit to occur 4 weeks after the last dose of study treatment) and Follow-up phase (8 weeks after the last dose of study treatment). Ongoing safety evaluation during Part 1 and Part 2 will be overseen by the Safety Evaluation Team (SET). In Part 3, ongoing safety and efficacy evaluation will be performed by the Independent Data Monitoring Committee (IDMC).

ELIGIBILITY:
Inclusion Criteria:

* Have received at least 3 prior lines of therapy including a proteasome inhibitor (PI) and an immunomodulatory agent (IMiD) in any order during the course of treatment for multiple myeloma or have disease that is refractory to both a PI and an IMiD
* Evidence of a response (partial response [PR] or better based on investigator's determination of response by International Myeloma Working Group [IMWG] criteria) to at least 1 prior treatment regimen
* Documented measurable disease for multiple myeloma at screening as defined in protocol
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies

Exclusion Criteria:

* Received any of the following prescribed medications or therapies in the past: Anti-CD38 antibody, including daratumumab, and/or Anti-PD-1 (programmed death-1) and anti-PD-L1 (programmed death-ligand 1) antibodies
* Plans to undergo a stem cell transplant prior to progression of disease on this study (these participants should not be enrolled to reduce disease burden prior to transplant)
* History of malignancy (other than multiple myeloma) within 2 years prior to first administration of study drug (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years)
* Clinical signs of meningeal involvement of multiple myeloma
* Known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal or known moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (13):
- Belgium (7):
  - ZNA Stuivenberg, Antwerp
  - Algemeen Ziekenhuis Klina, Brasschaat
  - AZ St.-Jan Brugge-Oostende AV, Bruges
  - UZBrussel, Brussels
  - UZA, Edegem
  - UZ Gent, Ghent
  - Az Groeninge, Kortrijk
- Israel (4):
  - Rambam Medical Center, Haifa
  - Carmel Hospital, Haifa
  - Hadassah Medical Center, Jerusalem
  - Sourasky Medical Center, Tel Aviv
- Spain (2):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Clinica Univ. de Navarra, Pamplona

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 10 participants were enrolled in the study. Among these, 9 participants were included in the Safety Run-in phase (Part 1) who received daratumumab intravenous (IV) and JNJ-63723283 IV and 1 participant randomized to Arm A in Part 2 of the study who received daratumumab IV alone.
Groups:
- Part 1: Daratumumab + JNJ-63723283: Participants in Safety Run-in cohort received daratumumab 16 mg/kg IV once every week (Weeks 1 to 8); then once every other week for 16 weeks (Weeks 9 to 24); then once every 4 weeks (Week 25 onwards) and JNJ-63723283 240 mg IV during Week 1 on Cycle 1 Day 2, Cycle 1 Day 15, then every 2 weeks thereafter. Each treatment cycle consisted of 28 days. Participants continued to receive study treatment until confirmed disease progression, unacceptable toxicity, or any other treatment discontinuation criteria were met.
- Part 2: Daratumumab (Arm A): Participants in treatment Arm A received daratumumab 16 mg/kg IV once every week (Weeks 1 to 8); then once every other week for 16 weeks (Weeks 9 to 24); then once every 4 weeks (Week 25 onwards). All participants were continued to receive study treatment until confirmed disease progression, unacceptable toxicity, or any other treatment discontinuation criteria were met.
Period: Overall Study
Arm/Group | Part 1: Daratumumab + JNJ-63723283 | Part 2: Daratumumab (Arm A)
Started | 9 | 1
Completed | 0 | 0
Not Completed | 9 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Sponsor Decision | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Daratumumab + JNJ-63723283 | Part 2: Daratumumab (Arm A) | Total
Number analyzed (Participants) | 9 | 1 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (10.97) | 43 | 61 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 1 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 1 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 4 | 0 | 4
  Israel | 4 | 1 | 5
  Spain | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) in Safety run-in Phase (Part 1)
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are adverse events (AEs) which will occur up to 2 years that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Up to 2 years
Population: Safety analysis set included all participants who have received at least 1 dose of study agent (JNJ-63723283 or daratumumab, partial or complete) in safety run-in phase of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Daratumumab + JNJ-63723283
Number analyzed (Participants) | 9
Participants | 9

2. Primary Outcome: Number of Participants With Dose Limiting Toxicity in Safety run-in Phase (Part 1)
Description: Dose limiting toxicity defined as an adverse event or adverse drug reaction experienced by the participants during observation of 28 days (Part 1) of treatment Cycle 1.
Time Frame: Cycle 1 (28 days)
Population: Safety analysis set included all participants who have received at least 1 dose of study agent (JNJ-63723283 or daratumumab, partial or complete) in safety run-in phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Daratumumab + JNJ-63723283
Number analyzed (Participants) | 9
Participants | 0

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) in Part 2
Description: as for outcome 1
Time Frame: Up to 2 years
Population: Safety analysis set included all participants who have received at least 1 dose of study agent in Part 2 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Daratumumab (Arm A)
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Part 1: Daratumumab + JNJ-63723283 | Part 2: Daratumumab (Arm A)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/1
Serious Adverse Events (participants affected / at risk) | 3/9 | 0/1
Other Adverse Events (participants affected / at risk) | 9/9 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Daratumumab + JNJ-63723283 (N=9) | Part 2: Daratumumab (Arm A) (N=1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Encephalitis Autoimmune (Nervous system disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Daratumumab + JNJ-63723283 (N=9) | Part 2: Daratumumab (Arm A) (N=1)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Corneal Degeneration (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Asthenia (General disorders) | 2 | 0
Chills (General disorders) | 2 | 0
Fatigue (General disorders) | 3 | 0
Influenza Like Illness (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Body Tinea (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Herpes Simplex (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Vulvovaginal Candidiasis (Infections and infestations) | 1 | 0
Lipase Increased (Investigations) | 1 | 0
Weight Decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Folate Deficiency (Metabolism and nutrition disorders) | 1 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Single participant enrolled in Part 2 was not evaluable for efficacy, hence data for Part 2 efficacy outcome measures was not collected. Sponsor suspended enrollment during Part 2, hence Part 2 stopped early, and Part 3 was not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT03357952/Prot_001.pdf
  • Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT03357952/SAP_000.pdf